CLINICAL TRIAL: NCT01370174
Title: Intervention to Enhance Lateral Balance Function and Prevent Falls in Aging
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Northwestern University (Other); VA Maryland Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vicki Gray, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: HP-00045644
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-06

CONDITIONS: Accidental Falls
Keywords: Falls; Balance; Protective Stepping; Lateral Balance; Elderly

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Induced Step Training (IST) (Active Comparator): The IST group will receive waist-pulls in both the left and right lateral directions by a motorized pulling system to produce stepping.
  Interventions: Other: Physical Training Interventions
- Hip Strength Training (HST) (Active Comparator): The HST group will have muscle strength training, to include hip abduction (AB) and adduction (AD) resistance exercises.
  Interventions: Other: Physical Training Interventions
- Combined Induced Step and Hip Strength Training (Active Comparator): This training group consists of combined induced step training (IST) and hip AB-AD strength training (HST).
  Interventions: Other: Physical Training Interventions
- Standard Flexibility and Relaxation (SFR) (Placebo Comparator): The SFR group will perform a flexibility and relaxation program involving minimal-intensity exercises.
  Interventions: Other: Physical Training Interventions

INTERVENTIONS:
Other: Physical Training Interventions — Subjects will be assigned to one of four training groups. Training will occur three times weekly for twelve consecutive weeks. The IST group will receive waist-pulls by a motorized machine to produce stepping. Subjects in the HST group will perform muscle resistance exercises. Subjects in the combined IST and HST will receive both IST and HST interventions. Participants in the SFR group will perform flexibility and relaxation exercises.

SUMMARY:
Falls and their consequences are among the major problems in the medical care of older individuals. The long-term goal of this research is to establish the efficacy of a scientifically grounded and mechanism-based therapeutic intervention for improving balance function and preventing falls in older people. When human balance is challenged, protective stepping is a vital strategy for preventing a fall during activities of daily life. Many older people at risk for falls have particular difficulties with successfully stepping sideways as a protective response to loss of balance in the lateral direction. We propose that age-related declines in lateral balance function through impaired protective stepping that precipitates falls, result from neuromechanical (NM) limitations in hip abductor-adductor (AB-AD) muscle strength (torque and power). Moreover, we hypothesize that these functional and NM impairments are reversible with combined high intensity induced step training (IST) and muscle strengthening.

DETAILED DESCRIPTION:
Falls and their consequences are among the major problems in the medical care of older individuals. Some 30 percent of community dwelling people aged 65 years and older, and over 50 percent of those living in institutions fall each year. Among older adults, complications of falls are the leading cause of deaths due to injury and are the most common cause of nonfatal injuries and hospitalization for trauma. The total lifetime healthcare cost of fall-related injuries for the elderly have been projected to reach $85 billion by the year 2020. Even in the absence of injury due to falling, the tendency to lose balance among the elderly commonly results in an overall reduction in the level of physical activity, and to a decreased ability to satisfactorily function in social roles.

Despite the contributions of multiple risk factors to age-related falls (e.g., environmental hazards, orthostatic hypotension, disorientation, sedation), it is well recognized that those who fall present greater impairments in neuromechanical (NM) factors than do older non-fallers. Aging changes in balance and gait associated with NM impairments have also been consistently found to be among the most important risk factors for falls. What is presently unresolved, however, is which among the age-associated NM impairments, altered balance and mobility functions are best associated with falls and responsive to interventions (training).

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Body Mass Index in range of 18.5 to 30

Exclusion Criteria:

* Timed -Up-and-Go faster than 12 seconds (very low fall risk)
* Persons advised by their doctor not to exercise
* Evidence of any medical condition as determined by physician or results of blood test that would lead to increased risk of accident, injury or illness due to any aspect of proposed tests and interventions, including resistance training
* Persons with history of brain, nerve or muscle disorder including Parkinson's disease, stroke, peripheral neuropathy or myopathy
* Persons with reported hip or knee joint replacement in past 6 months
* Persons with significant foot deformities or amputation as determined by a qualified medical professional
* Persons with sedative medications including hypnotics, anxiolytic, opioids, neuroleptics, or sedating antidepressants
* Persons using medications that pose a significant bleeding risks as determined by a qualified medical professional
* Any significant functional limitation as determined by a score of zero on any of the six daily tasks of the Instrumental Activities of Daily Living Scale (IADL) that enable independent living in the community. The six functional items used are: A. Telephone, B. Shopping, C. Food Preparation, D. Housekeeping, E. Laundry, and F. Transportation
* Non-ambulatory (unable to walk)
* Persons using a gait device at all times in home environment
* Cognitive impairment defined as Mini-Mental State Exam score <24
* Persons with uncorrected vision limiting visual function or eye surgery in ast 6 months
* Persons with uncorrected hearing impairment limiting daily activities or communication as determined by a qualified medical professional
* Persons with major depression (Centers for Epidemiological Studies Depression Survey score >16)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-01-25 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2017-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Rogers, PT, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - PTRS Research Lab, Baltimore, Maryland
  - VA Maryland Health Care System, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Induced Step Training (IST) | Hip Strength Training (HST) | Combined Induced Step and Hip Strength Training | Standard Flexibility and Relaxation (SFR)
Started | 25 | 26 | 25 | 26
Completed | 18 | 15 | 13 | 17
Not Completed | 7 | 11 | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Induced Step Training (IST) | Hip Strength Training (HST) | Combined Induced Step and Hip Strength Training | Standard Flexibility and Relaxation (SFR) | Total
Number analyzed (Participants) | 25 | 26 | 25 | 26 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 25 | 26 | 25 | 26 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (6.3) | 71.9 (6.8) | 73.3 (5.9) | 71.2 (4.2) | 72.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 11 | 18 | 61
  Male | 9 | 10 | 14 | 8 | 41
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 25 | 26 | 102

OUTCOME MEASURES:

1. Primary Outcome: Hip Abductor Torque
Description: Hip abductor torque at baseline and 3 months
Time Frame: At baseline and post-test at 3 months
Measure: Mean (Standard Error); unit: Nm/kg-m
Arm/Group | Induced Step Training (IST) | Hip Strength Training (HST) | Combined Induced Step and Hip Strength Training | Standard Flexibility and Relaxation (SFR)
Number analyzed (Participants) | 25 | 26 | 25 | 26
Nm/kg-m
  Baseline (Hip Strength Torque/Power) | 0.49 (0.04) | 0.49 (0.02) | 0.59 (0.04) | 0.0523 (0.03)
  Post-Test (Hip Strength Torque/Power) | 0.52 (0.03) | 0.61 (0.03) | 0.62 (0.05) | 0.55 (0.03)

2. Primary Outcome: Step Count
Description: The number of balance recovery steps at balance tolerance threshold at baseline and 3 months
Time Frame: At baseline and post-test at 3 months
Measure: Mean (Standard Error); unit: steps
Arm/Group | Induced Step Training (IST) | Hip Strength Training (HST) | Combined Induced Step and Hip Strength Training | Standard Flexibility and Relaxation (SFR)
Number analyzed (Participants) | 25 | 26 | 25 | 26
steps
  Baseline Balance Recovery Steps | 1.63 (.057) | 1.55 (.042) | 1.67 (.073) | 1.78 (.065)
  Post-Test Balance Recovery Steps | 1.14 (.080) | 1.24 (.12) | 0.97 (.067) | 1.24 (.099)

3. Secondary Outcome: Falls
Description: Analysis of fall history between falls in the year prior to enrollment and 12 months after training finished.
Time Frame: Individual subject at 12 months post training
Population: Not all study participants completed the falls following. The falls follow up was removed late in the trial.
Measure: Mean (95% Confidence Interval); unit: #falls/person/year
Arm/Group | Induced Step Training (IST) | Hip Strength Training (HST) | Combined Induced Step and Hip Strength Training | Standard Flexibility and Relaxation (SFR)
Number analyzed (Participants) | 18 | 15 | 13 | 17
#falls/person/year | 0.39 [0.19 to 00.82] | 0.27 [0.10 to 0.71] | 0.23 [0.07 to 0.72] | 0.88 [0.53 to 1.16]

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Induced Step Training (IST) | Hip Strength Training (HST) | Combined Induced Step and Hip Strength Training | Standard Flexibility and Relaxation (SFR)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 6/25 | 4/26 | 5/25 | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induced Step Training (IST) (N=25) | Hip Strength Training (HST) (N=26) | Combined Induced Step and Hip Strength Training (N=25) | Standard Flexibility and Relaxation (SFR) (N=26)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
R Leg Bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Fall (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Quad and Hip Abductor Soreness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
R Knee Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
R Arm Abrasion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Redness/Swelling of Scrotum (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Belching/Burping (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Muscle Soreness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hip Flexor Cramping (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Abdominal Cramping (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No